CLINICAL TRIAL: NCT01706653
Title: Fruit Polyphenols: Maximising Knowledge of Their Metabolic Health Benefits and Practical Applications
Brief Title: The Effects of a Polyphenol-enriched Fruit Drink on Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Lucozade Ribena Suntory (Industry)
Responsible Party: Principal Investigator, Dr Wendy Hall, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TSB101118; 12681-83204 (Other Grant/Funding Number: Technology Strategy Board)
Record Dates: First submitted 2012-10-10; First posted 2012-10-15 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Healthy Men and Women
Keywords: Polyphenol; Fruit; Metabolic; Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention 1 (Active Comparator): Polyphenol-enriched fruit-based drink - low
  Interventions: Dietary Supplement: Polyphenol-enriched fruit-based drink - low
- Intervention 2 (Active Comparator): Polyphenol-enriched fruit-based drink - medium
  Interventions: Dietary Supplement: Polyphenol-enriched fruit-based drink - medium
- Intervention 3 (Active Comparator): Polyphenol-enriched fruit-based drink - high
  Interventions: Dietary Supplement: Polyphenol-enriched fruit-based drink - high
- Intervention 4 (Placebo Comparator): Very low polyphenol fruit based drink (control)
  Interventions: Dietary Supplement: Very low polyphenol fruit based drink (control)

INTERVENTIONS:
Dietary Supplement: Polyphenol-enriched fruit-based drink - low
  Arms: Intervention 1
Dietary Supplement: Polyphenol-enriched fruit-based drink - medium
  Arms: Intervention 2
Dietary Supplement: Polyphenol-enriched fruit-based drink - high
  Arms: Intervention 3
Dietary Supplement: Very low polyphenol fruit based drink (control)
  Arms: Intervention 4

SUMMARY:
The purpose of this study is to determine whether consumption of the active product affects postprandial changes in metabolic indices, in comparison to the control product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living men aged from 20 to 60 years old, and postmenopausal women aged from 45 to 60 years old, on the day of inclusion
* Able to understand the information sheet and comply with all the trial procedures
* Having given written consent to take part in the study prior to participation.
* Body mass index (BMI): 18.0 - 35 kg/m².

Exclusion Criteria:

* Those diagnosed with Phenylketonuria (PKU)
* Those with known or suspected food intolerances, allergies or hypersensitivity
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study
* Women who are breast feeding
* Participation in another clinical trial
* Those who have donated blood within 3 months of the screening visit and participants for whom participation in this study would result in having donated more than 1500 millilitres of blood in the previous 12 months
* Those with Full Blood Counts and Liver Function test results outside of the normal range
* Pre-menopausal women due to the potential influence of cyclical changes in reproductive hormones on insulin sensitivity
* Current smokers, or reported giving up smoking within the last 6 months
* History of substance abuse or alcoholism
* Reported history of CVD, diabetes (or fasting glucose ≥ 7.1 mmol/L), cancer, kidney, liver or bowel disease, gastrointestinal disorder or use of drug likely to alter gastrointestinal function
* Unwilling to restrict consumption of specified high polyphenol foods for 24 h before the study
* Weight loss >3kg in preceding 2 months and body mass index <18 or >35 kg/m²
* Blood pressure ≥160/100 mmHg
* Total cholesterol ≥ 7.5 mmol/L; fasting triacylglycerol concentrations ≥ 5.0 mmol/L
* Medications that may interfere with the study such as alpha-glucosidase inhibitors (e.g. acarbose), insulin-sensitising drugs (e.g. metformin, thiazolidinediones), sulfonylureas, and lipid-lowering drugs. Other medications, should be reviewed by medical representative from KCL on a case by case basis.
* Nutritional supplements that may interfere with the study such as higher dose vitamins/minerals (>200% RNI), B vitamins, Vitamin C, calcium, copper, chromium, iodine, iron, magnesium, manganese, phosphorus, potassium and zinc. Subjects already taking vitamin or minerals at a dose around 100 % or less up to 200% of the RNI, or evening primrose/algal/fish oil supplements will be asked to maintain habitual intake patterns, ensuring that they take them every day and not sporadically. They will be advised not to stop taking supplements or start taking new supplements during the course of the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes & Nutritional Sciences Division, School of Medicine, King's College London, London, United Kingdom

REFERENCES:
- [Derived] Castro-Acosta ML, Smith L, Miller RJ, McCarthy DI, Farrimond JA, Hall WL. Drinks containing anthocyanin-rich blackcurrant extract decrease postprandial blood glucose, insulin and incretin concentrations. J Nutr Biochem. 2016 Dec;38:154-161. doi: 10.1016/j.jnutbio.2016.09.002. Epub 2016 Sep 14. PMID 27764725
- See also: Primary publication — http://www.ncbi.nlm.nih.gov/pubmed/27764725